CLINICAL TRIAL: NCT05409976
Title: Evaluation of the GORE® VIAFORT Vascular Stent for Treatment of Symptomatic Inferior Vena Cava Obstruction With or Without Combined Iliofemoral Obstruction
Brief Title: The GORE® VIABAHN® FORTEGRA Venous Stent IVC Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VNS 21-05
Record Dates: First submitted 2022-05-17; First posted 2022-06-08 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Venous Thromboses; Venous Disease; Venous Leg Ulcer; Venous Stasis; Venous Ulcer; Venous Stenosis; Venous Occlusion; Vein Thrombosis; Vein Occlusion; Vein Disease
Keywords: VIAFORT; Vein Stent; Venous Thrombosis; Venous Stenosis; Gore; Venous occlusion; VIABAHN FORTEGRA; FORTEGRA; Venous Disease; Deep Venous Insufficiency; Deep venous; DVT Treatment; Venous Stent; Venous insufficiency treatment options; Venous disease treatment Options
MeSH Terms: conditions — Venous Thrombosis; Varicose Ulcer

STUDY DESIGN:
Intervention Model Description: This study is a prospective, multicenter, non-randomized, single-arm study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- GORE® VIAFORT Vascular Stent (Experimental): GORE® VIAFORT Vascular Stent
  Interventions: Device: GORE® VIAFORT Vascular Stent

INTERVENTIONS:
Device: GORE® VIAFORT Vascular Stent — Treatment of symptomatic IVC obstruction with or without combined iliofemoral obstruction with the GORE® VIAFORT Vascular Stent.

SUMMARY:
This study is a prospective, multicenter, non-randomized, single-arm study to evaluate the performance, safety, and efficacy of the GORE® VIABAHN® FORTEGRA Venous Stent (formerly known as GORE® VIAFORT Vascular Stent) for treatment of symptomatic inferior vena cava obstruction with or without combined iliofemoral obstruction in adult patients.

DETAILED DESCRIPTION:
A maximum of 35 clinical investigative sites across the U.S., Europe, Australia, and New Zealand will participate in this study. One hundred and eleven subjects are intended to be implanted with the GORE® VIABAHN® FORTEGRA Venous Stent (formerly known as GORE® VIAFORT Vascular Stent) in this study, with a limit of 22 treated subjects per site and a minimum of 45 patients treated within the United States. Subjects will be evaluated through hospital discharge and return for follow-up visits at 1, 6, 12, 24, 36, 48, and 60 months post-treatment.

ELIGIBILITY:
Preoperative Inclusion Criteria:

* Patient is at least 18 years of age.
* Patient is willing and able to comply with all follow-up evaluations as well as any required medication or compression regimen.
* Patient is able to provide informed consent.
* One of the following: Clinical severity class of CEAP 'C' classification ≥3 or rVCSS pain score ≥2.
* Intention to treat the target areas with only the GORE® VIAFORT Vascular Stent.
* Estimated life expectancy ≥1 year.
* Patient is ambulatory (use of assistive walking device such as a cane or walker is acceptable).
* Patient has adequate inflow to the target lesion(s), per investigator/sub-investigator discretion, involving at least a patent femoral or deep femoral vein.

Preoperative Exclusion Criteria:

* Patient is a pregnant or breastfeeding woman, a woman planning to become pregnant through the 12-month visit, or a woman who is unwilling to practice an acceptable method of preventing pregnancy through the 12-month visit.
* Patient has clinically significant (e.g., symptoms of chest pain, hemoptysis, dyspnea, hypoxia, etc.) pulmonary embolism (confirmed via Computed Tomography Angiography) at the time of enrollment.
* Patient has a known uncorrectable bleeding diathesis or active coagulopathy meeting the following definitions: uncorrected INR>2 (not as a result of warfarin or DOAC therapy), OR platelet count <50,000 or >1,000,000 cells/mm3, OR white blood cell count <3,000 or >12,500 cells/mm3.
* Patient has impaired renal function (eGFR <30 mL/min/1.73m2) or is currently on dialysis.
* Patient has uncorrected hemoglobin of <9 g/dL.
* Patient has known history of antiphospholipid syndrome (APS) or patients with hypercoagulable states that are unwilling to take anticoagulant medications on a long-term basis.
* Patient has known homozygous inherited coagulation defect or Protein C/S deficiency.
* Patient has a planned surgical intervention (other than pre-stenting procedures such as thrombolysis or thrombectomy) within 30 days prior to or within 30 days after the planned study procedure.
* Patient is currently participating in another investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the endpoints of this treatment, in the opinion of the investigator/sub-investigator. Observational studies are permitted.
* Patient has had a previous major (i.e., above the ankle) amputation of the target lower limb.
* Patient has known sensitivity to device materials or contraindication to antiplatelets, thrombolytics, anticoagulants (including patients with known prior instances of Heparin Induced Thrombocytopenia type 2 (HIT-2)), or iodinated contrast.
* Patient has had prior stenting or grafts in the target vessels.
* Patient has a known or suspected active systemic infection at the time of the index procedure. Patients with a chronic infection (e.g., HIV, hepatitis C) that is well controlled under their current treatment regimen may be eligible.
* Patient has known history of intravenous drug abuse within one year of treatment.
* Patient has significant peripheral arterial disease (chronic Rutherford Type 2 or greater, acute Rutherford Type IIa or greater).
* Patient has a BMI >40.
* Patient is actively undergoing or plans to begin cancer treatment.

Intraoperative Inclusion Criteria:

* Presence of non-malignant obstruction of the inferior vena cava defined as occlusion or at least 50% reduction in target vessel lumen as measured by procedural IVUS and venogram, with or without non-malignant obstruction of the common femoral vein, external iliac vein, and/or common iliac vein.
* Patient can accommodate an appropriately sized GORE® VIAFORT Vascular Stent as per reference vessel diameter (see IFU), as determined by intraoperative IVUS post pre-dilation.
* Patient must have appropriate access vessels to accommodate the delivery sheath for the selected device size.
* Patient has adequate landing zones free from significant disease requiring treatment within the native vessels beyond the proximal and distal margins of the lesion.
* Patient has adequate inflow to the target lesion(s), per investigator/sub-investigator discretion, involving at least a patent femoral or deep femoral vein.
* Lesion can be traversed with a guidewire.
* Disease involves the inferior vena cava and may include iliofemoral segments with intent to stent all affected iliofemoral and caval segments.
* Patient does not have significant (i.e., >20% residual thrombosis) acute thrombus within the target stent area at the time of investigational device placement. Patients with acute thrombus within the target stent area must have thrombus successfully treated prior to investigational device placement. Successful thrombus treatment is defined as reestablishment of antegrade flow with ≤20% residual thrombosis as confirmed by IVUS and venogram, AND freedom from bleeding, vascular injury, or hemodynamically significant pulmonary embolism. After successful thrombus treatment, investigational device placement can occur within the same procedure.
* Patient does not have an inferior vena cava filter present within the target stent area at the time of investigational device placement. Patients with an inferior vena cava filter present within the target stent area must have the filter successfully removed prior to investigational device placement. Successful removal is defined as removal of the main body of the filter and intra-luminal fragments such that there is minimal risk to luminal integrity per investigator/sub-investigator discretion AND freedom from bleeding, vascular injury, or hemodynamically significant pulmonary embolism. After successful filter removal, investigational device placement can occur within the same procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2022-10-25 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Composite of efficacy and safety events | 12 months
  Composite primary endpoint consisting of freedom from the following:
  * Loss of primary patency through 12-month follow-up
  * Stent embolization through 12-month follow-up
  * Device- or procedure-related death through 30 days
  * Clinically significant pulmonary embolism confirmed via Computed Tomography Angiography through 30 days
  * Device- or procedure-related vascular injury through 30 days requiring surgical or endovascular intervention
  * Device- or procedure-related major bleeding events through 30 days

SECONDARY OUTCOMES:
Number of subjects with primary patency as confirmed by imaging and adverse events | 60 months
  Number of subjects with freedom from both:
  * stent occlusion due to restenosis or thrombosis as confirmed with imaging, and
  * clinically driven target lesion revascularization as confirmed with imaging and adverse events
Number of subjects with secondary patency as confirmed by imaging and adverse events | 60 months
  Number of subjects with freedom from permanent loss of blood flow through the device, regardless of reintervention.
Number of subjects with clinically driven target lesion revascularization as confirmed by imaging and adverse events | 60 months
  Number of subjects with repeat endovascular procedures (e.g., PTA, stenting, thrombectomy/thrombolysis) to restore flow, performed within the margins of the investigational devices due to ≥50% restenosis of the target lesion as measured via imaging AND the failure to improve or recurrence of venous origin leg pain or venous edema related to the target lesion present at baseline, or the onset of new symptoms including venous origin pain and venous edema related to the target lesion.
Number of subjects with device fracture as confirmed with imaging | 60 months
  Number of subjects with device fracture as confirmed with imaging.
Number of subjects with stent embolization as confirmed with imaging | 12 months
  Number of subjects with stent embolization as confirmed with imaging.
Number of subjects with device- or procedure-related death | 30 days
  Number of subjects with device- or procedure-related death.
Number of subjects with clinically significant pulmonary embolism as confirmed with imaging and adverse events | 30 days
  Number of subjects with clinically significant pulmonary embolism confirmed via Computed Tomography Angiography through 30 days.
Number of subjects with device- or procedure-related vascular injury as confirmed with adverse events | 30 days
  Number of subjects with device- or procedure-related vascular injury through 30 days requiring surgical or endovascular intervention.
Number of subjects with device- or procedure-related major bleeding events as confirmed with adverse events | 30 days
  Number of subjects with device- or procedure-related major bleeding events through 30 days.
Revised Venous Clinical Severity Scale (rVCSS) | 60 months
  Change in Revised Venous Clinical Severity Scale (rVCSS) Measurement through 60-month follow-up compared to baseline prior to treatment.
  Note: The rVCSS scale ranges from 0 to 30, with higher scores reflecting worse symptoms.
Revised Venous Clinical Severity Scale (rVCSS) Pain | 60 months
  Change in Revised Venous Clinical Severity Scale (rVCSS) Pain Measurement through 60-month follow-up compared to baseline prior to treatment.
  Note: The rVCSS Pain scale ranges from 0 to 3, with higher scores reflecting worse pain.
Venous Insufficiency Epidemiological and Economic Study - Quality of Life/Symptoms (VEINES-QOL/Sym) VEINES-QOL/Sym | 60 months
  Change in Venous Insufficiency Epidemiological and Economic Study - Quality of Life/Symptoms (VEINES-QOL/Sym) Measurement through 60-month follow-up compared to baseline prior to treatment.
Villalta | 60 months
  Change in Villalta Measurement through 60-month follow-up compared to baseline prior to treatment.
5 Level EuroQol-5 Dimension (EQ-5D-5L) | 60 months
  Change in 5 Level EuroQol-5 Dimension (EQ-5D-5L) Measurement through 60-month follow-up compared to baseline prior to treatment.
Technical success | Index procedure (post-op day 0)
  Number of subjects with successful delivery and deployment of the stent to the intended location, and removal of delivery system.
Lesion success | Index procedure (post-op day 0)
  Number of subjects with evidence of ≤50% residual stenosis at the conclusion of the index procedure as measured by IVUS or venogram.
Procedural success | Index procedure through hospital discharge (discharge estimated as up to 30 days post-treatment)
  Number of subjects with lesion success and the absence of major adverse events (i.e., stent embolization, device- or procedure-related death, clinically significant pulmonary embolism, device- or procedure-related vascular injury requiring surgical or endovascular intervention, and device- or procedure-related major bleeding) prior to discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Kush Desai, MD, Principal Investigator — Northwestern University; Stephen Black, MD, FRCS (Ed), FEBVS, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (17):
- United States (8):
  - Stanford University School of Medicine, Stanford, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Northwestern, Chicago, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - Mount Sinai Medical Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Atrium Health-Sanger Heart and Vascular Institute, Charlotte, North Carolina
  - Sentara, Norfolk, Virginia
- Flinders Medical Centre, Adelaide, South Australia, Australia
- Germany (2):
  - Universitätsklinikum Aachen, Aachen
  - Alexianer Klinikum Hochsauerland GmbH, Arnsberg
- University College Hospital GALWAY /Clinical Research Facility Galway, Galway, Connacht, Ireland
- Italy (2):
  - Ospedale San Raffaele, Milan
  - Hesperia Hospital, Modena
- Auckland City Hospital, Auckland, New Zealand
- United Kingdom (2):
  - Addenbrooke's Hospital, Cambridge
  - St Thomas' Hospital, London

IPD SHARING:
Plan to Share IPD: No